CLINICAL TRIAL: NCT01941667
Title: Transitional Telehealth Home Care: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-008246
Record Dates: First submitted 2013-02-28; First posted 2013-09-13 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Congenital Heart Disease; Post Cardiac Surgery
Keywords: Congenital Heart Disease; Neonates and infants; Telehealth; Virtual Home Visits
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily Messages, virtual home visits (Experimental): Intervention includes: Measuring daily weights, 24 hour intake, heart rate, oxygen level
  Daily messages requesting weight, intake, pulse ox and pulse are automated
  Virtual home visits occur twice weekly where the investigators see the infant and families.
  Interventions: Behavioral: Daily Messages, Virtual Home Visits
- Usual Care (Placebo Comparator): Infants will have usual care as defined by cardiology.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Daily Messages, Virtual Home Visits — Intervention includes: Measuring daily weights, 24 hour intake, heart rate, oxygen level
  Daily messages requesting weight, intake, pulse ox and pulse are automated
  Virtual home visits occur twice weekly where the investigators see the infant and families.
  Arms: Daily Messages, virtual home visits
Other: Usual Care — Usual care as defined by by the Cardiology Department.
  Arms: Usual Care

SUMMARY:
The investigators want to determine if additional, increased contact with infants and families discharged to home after cardiac surgery improves infant and parent outcomes as compared to usual care.

DETAILED DESCRIPTION:
The investigators want to compare videoconferencing (SKYPE or FACTIME) and a monitoring system called Buddy Check is helpful. Buddy Check is a web-based tool using speech and internet technology to maintain contact with the health care team.

Infants are randomized to usual care or the intervention which uses automated daily phone calls and 2 virtual home visits each week. Weights, oxygen levels, and amount of food taken are obtained by the primary caregiver (parent) daily and sent via automated phone call, text message or email messages based on primary caregiver's desired.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery within 2.5 weeks of life,
* Diagnosis of congenital heart disease,
* Post menstrual age 37 weeks and older;
* Minimum birth weight 2500 grams,
* At least one parent speaks and reads English,
* Anticipated discharge by 21 days of life

Exclusion Criteria:

* Cardiomyopathy,
* Diagnosis of Genetic syndrome

Ages: 2 Weeks to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2012-07; Primary Completion 2016-11 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Parental Stress Score | Within 5 months of infant's life
  Parental Stress will be measured through the use of the total score of Parental Stress Index collected at the completion of the study period for the infant and family, approximately 5 months of infant's life.

SECONDARY OUTCOMES:
Parental Quality of life Score | Within 5 months of infant's life
  Parental Quality of life will be measured by total score of "QOL, The Ulm Quality of Life Inventory for Parents (ULQIE)" collected at the completion of the study period for the infant and family, approximately 5 months of infant's life.
Parental Social Isolation Score | Within 5 months of Infant's life.
  Parental social isolation will be measured by the total score on the Enriched SocialSupport Index with higher scores indicating more support which is collected within 5 months of the infant's life.
Weight Gain at 5 months. | Within 5 months of life
  Weight gain will be measured by change in z scores of infant's weight (measured in grams)which will be obtained at discharge from the hospital and at the end of the study period, approximately 5 months of life.
Post Traumatic Stress Disorder Symptoms | Within 5 month's of Infant's Life
  Post Traumatic Stress Disorder Symptoms will be measured by the number of symptoms on the Post Traumatic Stress Disorder Scale at the end of the study period, within 5 months of the infant's life.

OTHER OUTCOMES:
Health Care Resource Utilization | Within 5 month's of infants life.
  Health Care Utilization will be measured by per patient costs based on number of re-hospitalizations, Length of Stay of re-hospitalization, number of emergency department visits and number of acute care visits within 5 months of infant's life.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Medoff-Cooper, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of PHiladelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lisanti AJ, Golfenshtein N, Min J, Medoff-Cooper B. Early growth trajectory is associated with psychological stress in parents of infants with congenital heart disease, but moderated by quality of partner relationship. J Pediatr Nurs. 2023 Mar-Apr;69:93-100. doi: 10.1016/j.pedn.2022.12.016. Epub 2023 Jan 23. PMID 36696826
- [Derived] Golfenshtein N, Lisanti AJ, Cui N, Cooper BM. Predictors of Post-traumatic stress symptomology in parents of infants with Congenital Heart Disease post-surgery and after four months. J Pediatr Nurs. 2022 Jan-Feb;62:17-22. doi: 10.1016/j.pedn.2021.11.013. Epub 2021 Nov 25. PMID 34839196
- [Derived] Medoff Cooper B, Marino BS, Fleck DA, Lisanti AJ, Golfenshtein N, Ravishankar C, Costello JM, Huang L, Hanlon AL, Curley MAQ. Telehealth Home Monitoring and Postcardiac Surgery for Congenital Heart Disease. Pediatrics. 2020 Sep;146(3):e20200531. doi: 10.1542/peds.2020-0531. PMID 32817266